CLINICAL TRIAL: NCT02919670
Title: A Randomized Double-Blinded Phase 2 Study Evaluating a Proprietary Amino Acid Mixture (Enterade®) in Patients Receiving High-Dose Melphalan Conditioning Followed by Autologous Stem Cell Transplantation for Multiple Myeloma and Non-Hodgkin Lymphoma
Brief Title: A Study Evaluating a Proprietary Amino Acid Mixture (Enterade®) in Patients Receiving High-Dose Melphalan Conditioning Followed by Autologous Stem Cell Transplantation for Multiple Myeloma and Non-Hodgkin Lymphoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Entrinsic Health (Unknown)
Responsible Party: Principal Investigator, Mahasweta Gooptu, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 16-329
Record Dates: First submitted 2016-09-26; First posted 2016-09-29 (Estimated); Results first posted 2023-03-16 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2022-06

CONDITIONS: Multiple Myeloma; Non-Hodgkin's Lymphoma
Keywords: Stem Cell Transplant
MeSH Terms: conditions — Multiple Myeloma; Lymphoma, Non-Hodgkin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Enterade and Standard Supportive Care (Experimental): * Two 8 oz. bottles of Enterade will be administered daily
  * Enterade will be given orally from admission until day +14 or until discharge
  * Standard Supportive Care will be administered according to institution's practice
  Interventions: Dietary Supplement: Enterade; Other: Standard Supportive Care
- Placebo and Standard Supportive Care (Placebo Comparator): * Two 8 oz. bottles of Placebo will be administered daily
  * Placebo will be given orally from admission until day +14 or until discharge
  * Standard Supportive Care will be administered according to institution's practice
  Interventions: Dietary Supplement: Placebo; Other: Standard Supportive Care

INTERVENTIONS:
Dietary Supplement: Enterade
  Arms: Enterade and Standard Supportive Care
Dietary Supplement: Placebo
  Arms: Placebo and Standard Supportive Care
Other: Standard Supportive Care

SUMMARY:
This research study is evaluating Enterade, a supplement, as a possible treatment for the side effects caused by Stem Cell Transplant.

The following interventions will be involved in this study:

* Enterade plus standard supportive care
* Placebo plus standard supportive care. The placebo will be a mixture of water, electrolytes, and sweetener.

DETAILED DESCRIPTION:
This research study is a Phase II clinical trial. Phase II clinical trials test the safety and effectiveness of an investigational intervention to learn whether the intervention works in treating a specific disease, or in this case, the side effects from a standard treatment for Stem Cell Transplant side effect. "Investigational" means that the intervention is being studied.

In this research study, the investigators are evaluating Enterade/Placebo plus standard supportive care for the treatment of the side effects caused by transplant. Enterade works by rehydrating the intestinal cells, thereby helping to restore normal bowel function. The ingredients in Enterade are generally recognized as safe by the Food and Drug Administration. This research study is hoping to learn if adding Enterade to the standard supportive care regimen for the participant transplant will help reduce the side effects from the transplant.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histologically or cytologically confirmed Multiple Myeloma, or Non-Hodgkin Lymphoma and must be undergoing Melphalan conditioning for autologous HSCT.
* Age equal or greater than 18 years old.
* ECOG performance status ≤2 (Karnofsky ≥60%)
* Participants must have adequate organ and marrow function to proceed to transplant.
* Ability to tolerate thin liquids by mouth at the time of admission.
* The effects of Enterade® on the developing human fetus are unknown. For this reason and other therapeutic agents used in this trial are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) at the time of study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of the trial.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Participants who have had radiotherapy within 4 weeks prior to entering the study or those who have not recovered from adverse events due to chemotherapy agents administered during this time period.
* Participants who are receiving any other investigational agents. Participants who are receiving standard of care induction therapy on a clinical trial may be eligible after discussion with the overall principal investigator.
* Participants with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
* Known allergy to Stevia.
* Participants receiving any medications or antibiotics to treat Clostridium difficile infection prior to the initiation of the study will be ineligible for this study.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active Clostridium difficile infection or history of Clostridium difficile infection.
* Participants with evidence of diarrhea as defined by three or more loose or liquid stools per day or loose watery stool (greater volume of stool), that occurs more frequently than usual and lasting for more than three days prior to admission, history of inflammatory bowel disease, irritable bowel syndrome, colectomy or bariatric surgery, Celiac disease.
* Participants with psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant and nursing women are excluded from this study because of teratogenicity and toxicity risks associated with the conditioning regimen for patients undergoing autologous HSCT.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2016-10; Primary Completion 2019-05 (Actual); Study Completion 2020-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mahasweta Gooptu, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 10/5/2016 - 10/05/2017
Pre-assignment Details: Of 114, 6 patients did not receive transplant and 1 patient had a delayed transplant..5 patients withdrew consent , 1 patient did not take any amount due to the finding mold, 1 patient did not take due to subjects inability to swallow liquids and 1 patient had an insurance issue. Thus a total of 15 patients are excluded. (114-15=99).
Groups:
- Enterade and Standard Supportive Care: * Two 8 oz. bottles of Enterade will be administered daily
  * Enterade will be given orally from admission until day +14 or until discharge
  * Standard Supportive Care will be administered according to institution's practice
  Enterade
  Standard Supportive Care
- Placebo and Standard Supportive Care: * Two 8 oz. bottles of Placebo will be administered daily
  * Placebo will be given orally from admission until day +14 or until discharge
  * Standard Supportive Care will be administered according to institution's practice
  Placebo
  Standard Supportive Care
Period: Overall Study
Arm/Group | Enterade and Standard Supportive Care | Placebo and Standard Supportive Care
Started | 49 | 50
Completed | 6 | 11
Not Completed | 43 | 39
Not completed — Only 17 participants met compliance | 43 | 39

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Enterade and Standard Supportive Care | Placebo and Standard Supportive Care | Total
Number analyzed (Participants) | 49 | 50 | 99
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 44 | 44 | 88
  >=65 years | 5 | 6 | 11
Age, Continuous [Median (Full Range); unit: years] | 61 [25 to 74] | 59 [40 to 77] | 60 [25 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 10 | 25
  Male | 34 | 40 | 74
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 4 | 7
  White | 45 | 44 | 89
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 49 | 50 | 99
Count of participants [Count of Participants; unit: Participants] | 49 | 50 | 99

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Grade 3 or Higher Diarrhea GI Toxicity
Description: Evaluation will made using Fisher's exact test. Among 99 participants who received some intervention
Time Frame: 14 days
Population: Only 17 participants met the protocol definition of compliance
Measure: Count of Participants; unit: Participants
Groups:
- Enterade: Participants who received Enterade
- Placebo: Participants who received placebo
Arm/Group | Enterade | Placebo
Number analyzed (Participants) | 49 | 50
Participants | 18 | 21

2. Secondary Outcome: Maximum Daily Stool Frequency
Time Frame: 14 days
Population: Only 17 participants met the protocol definition of compliance
Measure: Mean (Full Range); unit: number of stools per day
Groups:
- Enterade: Participants who took Enterade
- Placebo: Participants who took placebo
Arm/Group | Enterade | Placebo
Number analyzed (Participants) | 49 | 50
number of stools per day
  Day +1 to Day +7 | 5 [1 to 18] | 6 [1 to 30]
  Day +8 to Day +14 | 6 [0 to 34] | 5 [1 to 75]

3. Secondary Outcome: Percentage of Participants With Diarrhea on the Day of Maximum Daily Stool Frequency
Time Frame: 14 days
Population: Only 17 participants met the protocol definition of compliance
Measure: Count of Participants; unit: Participants
Arm/Group | Enterade | Placebo
Number analyzed (Participants) | 49 | 50
Participants
  Day +1 to Day +7 | 22 | 26
  Day +8 to Day +14 | 25 | 22

4. Secondary Outcome: Duration Of Hospitalization (Days) From Admission To Discharge
Time Frame: Up to 45 days
Population: Only 17 participants met the protocol definition of compliance
Measure: Median (Full Range); unit: days
Arm/Group | Enterade and Standard Supportive Care | Placebo and Standard Supportive Care
Number analyzed (Participants) | 49 | 50
days | 17 [14 to 29] | 17 [13 to 45]

5. Secondary Outcome: Percent Change in Weight From Baseline to Day 14
Time Frame: baseline and day 14
Population: Only 17 participants met the protocol definition of compliance
Measure: Median (Full Range); unit: percent change
Arm/Group | Enterade and Standard Supportive Care | Placebo and Standard Supportive Care
Number analyzed (Participants) | 49 | 50
percent change | -2.5 [-18.4 to 11.6] | -2.2 [-9 to 45.9]

6. Secondary Outcome: Median Amount Of Anti-Diarrheal Medications
Time Frame: 14 days
Measure: Median (Full Range); unit: mg
Arm/Group | Enterade and Standard Supportive Care | Placebo and Standard Supportive Care
Number analyzed (Participants) | 49 | 50
mg | 27 [2 to 264] | 30 [2 to 160]

7. Secondary Outcome: the Tolerability of Enterade® as Measured by the Number of Compliant Patients
Time Frame: 14 days
Population: Patients who take the study drug two 8 oz. bottles (480 ml) daily for at least 11 days are regarded as compliant. Compliance is assessed among patients who received any amount of the study drug (N=99).Only 17 participants met the protocol definition of compliance
Measure: Count of Participants; unit: Participants
Arm/Group | Enterade and Standard Supportive Care | Placebo and Standard Supportive Care
Number analyzed (Participants) | 49 | 50
Participants | 6 | 11

8. Secondary Outcome: Calorie Consumption
Time Frame: 14 days
Population: Only 17 participants met the protocol definition of compliance
Measure: Median (Full Range); unit: calories
Arm/Group | Enterade and Standard Supportive Care | Placebo and Standard Supportive Care
Number analyzed (Participants) | 49 | 50
calories
  Admission | 1848.5 [352 to 2919] | 1790 [680 to 2793]
  D+7 | 625.5 [0 to 2523] | 720 [0 to 2770]
  D+14 | 800 [0 to 2300] | 922 [0 to 3174]

9. Secondary Outcome: Number of Participants With Fever or Neutropenia
Time Frame: 14 days
Population: Only 17 participants met the protocol definition of compliance
Measure: Count of Participants; unit: Participants
Arm/Group | Enterade and Standard Supportive Care | Placebo and Standard Supportive Care
Number analyzed (Participants) | 49 | 50
Participants
  Fever | 3 | 3
  Neutrophil count decreased | 28 | 30

ADVERSE EVENTS:
Time Frame: 14 days
Description: The primary endpoint is the incidence of NCI-CTCAE 4.0 grade 3 or higher GI toxicity in the 14 days following autologous HSCT
Arm/Group | Enterade and Standard Supportive Care | Placebo and Standard Supportive Care
All-Cause Mortality (participants affected / at risk) | 0/49 | 1/50
Serious Adverse Events (participants affected / at risk) | 0/49 | 1/50
Other Adverse Events (participants affected / at risk) | 18/49 | 21/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Enterade and Standard Supportive Care (N=49) | Placebo and Standard Supportive Care (N=50)
Clostridium septicum septic shock (Infections and infestations) | NA | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Enterade and Standard Supportive Care (N=49) | Placebo and Standard Supportive Care (N=50)
Colitis (Infections and infestations) | 3 | 3
Diarrhea (Gastrointestinal disorders) | 7 | 12
Dysphagia (Gastrointestinal disorders) | 0 | 1
Esophagitis (Gastrointestinal disorders) | 2 | 5
Mucositis oral (Infections and infestations) | 4 | 0
Nausea (Gastrointestinal disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2019-05-06): https://cdn.clinicaltrials.gov/large-docs/70/NCT02919670/Prot_000.pdf
  • Statistical Analysis Plan (2017-04-26): https://cdn.clinicaltrials.gov/large-docs/70/NCT02919670/SAP_001.pdf